CLINICAL TRIAL: NCT05169398
Title: EUS-guided Hepatico-gastrostomy Using a Novel Lumen Apposing Metal Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2021.447
Record Dates: First submitted 2021-11-12; First posted 2021-12-27 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Malignant Biliary Obstruction
Keywords: Malignant Biliary Obstruction; EUS-biliary drainage; EUS-guided hepaticogastrostomy

STUDY DESIGN:
Intervention Model Description: EUS-guided hepaticogastrostomy would be performed with the MG-biliary stent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-guided hepaticogastrostomy (Experimental): EUS-guided hepaticogastrostomy would be performed with the MG-biliary stent (Niti-S, Taewoong Medical, Gyeonggi-do, Korea).
  Interventions: Device: EUS-guided hepaticogastrostomy

INTERVENTIONS:
Device: EUS-guided hepaticogastrostomy — EUS-guided hepaticogastrostomy would be performed with the MG-biliary stent (Niti-S, Taewoong Medical, Gyeonggi-do, Korea)

SUMMARY:
EUS-guided biliary drainage is gaining popularity as a means of achieving endoscopic drainage in patients with failed endoscopic retrograde cholangiopancreatography (ERCP) 1. EUS-guided hepaticogastrostomy (HGS) is a type of EUS-guided biliary drainage and the procedure is employed when the ERCP fails due to a malignant bile duct obstruction but the papilla is inaccessible or if the first of the duodenum is infiltrated by tumor. Recently, a novel dedicated HGS (Niti-S, Taewoong Medical, Gyeonggi-do, Korea) has become available, the stent has a novel design to that prevents the stent from migration, further improving the safety.

The aim of the current study is to evaluate the feasibility and outcomes of the novel lumen apposing stent for EUS-guided HGS. The hypothesis is that the device is safe and effective.

DETAILED DESCRIPTION:
This is a prospective feasibility study enrolling patients suffering from malignant biliary obstruction with failed or anticipated difficult ERCP. Consecutive patients satisfying the inclusion criteria would be recruited.

EUS-guided hepaticogastrostomy would be performed with the MG-biliary stent. The MG-biliary stent (Niti-S, Taewoong Medical, Gyeonggi-do, Korea) is a novel device designed for hepaticogastrostomy. The stent is a partially covered metal stent made by nitinol covered with silicone. One end of the stent is uncovered and designed for placement in the intrahepatic ducts. The other end has a self-folding design that creates a flange and prevents migration of the stent outside the stomach. The stent diameter is either 8 or 10mm and the length can be 6,8,10 or 12cm long.

Outcome parameters include safety, technical and clinical success

ELIGIBILITY:
Inclusion Criteria:

1. >= 18 years of age
2. Anatomically feasible for EUS-guided hepatico-gastrostomy
3. Patients with clinical symptoms and/or signs of extrahepatic biliary obstruction (jaundice, biliary-type pain, cholangitis)
4. Patients with unsuccessful ERCP (failed ERCP, anticipated difficult ERCP or high risk for pancreatitis)
5. Written informed consent (and assent when applicable) obtained from subject.

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Coagulopathic patients (INR>1.5, platelets <50,000)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event | 30 day
  a life-threatening or severe event requiring endoscopic and/or surgical intervention, transfusion or IV/IM antibiotics

SECONDARY OUTCOMES:
Number of patients with technical success | 1 day
  transmural placement of the stent across the stomach or duodenum into the bile duct
Number of patients with Clinical success | 7 days
  decrease of >20% bilirubin from baseline level
Stent patency | 1 year
  the period between stent insertion and stent occlusion or stent removal

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogura T, Ueno S, Okuda A, Nishioka N, Yamada M, Matsuno J, Ueshima K, Yamamoto Y, Higuchi K. Technical feasibility and safety of one-step deployment of EUS-guided hepaticogastrostomy using an 8-mm diameter metal stent with a fine-gauge stent delivery system (with video). Endosc Ultrasound. 2021 Sep-Oct;10(5):355-360. doi: 10.4103/EUS-D-20-00206. PMID 34427190
- [Result] Teoh AYB, Dhir V, Kida M, Yasuda I, Jin ZD, Seo DW, Almadi M, Ang TL, Hara K, Hilmi I, Itoi T, Lakhtakia S, Matsuda K, Pausawasdi N, Puri R, Tang RS, Wang HP, Yang AM, Hawes R, Varadarajulu S, Yasuda K, Ho LKY. Consensus guidelines on the optimal management in interventional EUS procedures: results from the Asian EUS group RAND/UCLA expert panel. Gut. 2018 Jul;67(7):1209-1228. doi: 10.1136/gutjnl-2017-314341. Epub 2018 Feb 20. PMID 29463614